CLINICAL TRIAL: NCT03836885
Title: The APOLP Trial: A Single-Center, Randomized, 16 Weeks, Explanatory, Parallel-Group, Superiority, Blinded, Placebo-Controlled, Clinical Trial of Apremilast Use in Oral Lichen Planus
Brief Title: Apremilast - Oral Lichen Planus Trial
Acronym: APOLP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to delay in enrollment.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Celgene (Industry); Sunnybrook Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Hagen Klieb, Oral Pathologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 049-2018
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apremilast (Experimental): Oral tablet
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator): Oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast tablets. Titration will occur in the initial five days of treatment as per dosing in psoriasis as follows: Day 1: 10 mg; Day 2: 20 mg; Day 3: 30 mg; Day 4: 40 mg; Day 5: 50 mg. Day 6 and thereafter patients will be dosed at 60 mg for a total of 12 weeks.
  Other Names: Otezla
  Arms: Apremilast
Drug: Placebo — Placebo Oral tablets. Patients randomized to the control arm will receive color, taste, shape and odour matched oral placebo. The number of tablets and the days taken is analogous to the intervention arm had they been randomized to the intervention arm.
  Arms: Placebo

SUMMARY:
Apremilast for the management of oral lichen planus.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) affects approximately 1.27% of the general population. Inflammatory responses constitute a major component of OLP pathogenesis where targeted therapies play an important role in managing this condition. Apremilast is a new well-tolerated and relatively safe anti-inflammatory therapy that has been approved for managing psoriasis and psoriatic arthritis. Given its safer profile, Apremilast may ameliorate inflammatory responses in clinically active OLP without the experience of serious adverse events associated with other systemic immunosuppressive therapies used to treat OLP. The plan is to conduct a single-center, explanatory, randomized, 16 weeks, parallel group, superiority, blinded, placebo-controlled, clinical trial.

The main objective is treatment success assessment. Other objectives include exploring the efficacy of Apremilast in clinically active OLP adult patients considered for systemic treatment and failed topical corticosteroid therapy. It is hypothesized that Apremilast will induce more treatment success as compared to placebo in patients who failed the standard treatment of topical corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to participate in this study:

1. Must be 18 years or older at time of consent.
2. Patients must have clinically active OLP that is being considered for systemic therapy; and an oral biopsy within the last 12 months of randomization showing a lichenoid reaction correlating clinically with OLP.
3. Must have failed topical corticosteroids therapy. Topical corticosteroid failure is defined as receiving a trial of at least 4 weeks of high potency topical corticosteroids without achieving sufficient improvement by patients.
4. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions). Laboratory work-up includes the following: complete blood count (CBC), creatinine, albumin, aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), total bilirubin, serum, Beta-HCG (if female), Hepatitis C antibodies and HgbA1C.
5. Male participants must use a recognized effective method of contraception with any female partner (i.e. at a minimum, barrier plus an additional method of contraception) while on investigational product and for at least 4 weeks after taking the last dose of investigational product.
6. Female participants of childbearing potential (FCBP)† must have a negative pregnancy test at Screening. While on investigational product and for at least 4 weeks after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below:

   1. Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; prior hysterectomy; prior bilateral oophorectomy or salpingo-oophorectomy; or partner's vasectomy;

      OR
   2. Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; plus one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

      * A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).
      * The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

Exclusion Criteria:

All participants meeting any of the following exclusion criteria at baseline will be excluded from participation in this study:

1. Inability to give written consent by the patient or alternative decision maker (will be assessed at screening visit).
2. Unwillingness to use at least one effective method of contraception due to unknown fetal risks
3. Use of systemic or topical therapy for OLP other than allowed concomitant care for symptomatic relief in the past 4 weeks.
4. Hypersensitivity to Apremilast or use of Apremilast within 4 weeks prior to start of study drug. The contraindications to Apremilast use include prior hypersensitivity reactions, breast-feeding, and pregnancy (Uptodate.com® accessed August 1st, 2016). An increased incidence of depression or depressed mood by 1.3% for Apremilast 30 mg BID (twice a day) (OTEZLA® drug monograph accessed August 1st, 2016) was observed in phase 3 psoriasis studies. Celgene suggests that prescribers should carefully weigh the risks and benefits in patients with a history of depression and/or suicidal thoughts or behaviour. The research team will discuss these psychiatric adverse events in the screening visit where patients/caregivers will be instructed to notify the treating team for any mood changes.
5. History of palpitations/tachyarrhythmia, severe renal impairment (eGFR less than or equal to 29), or lactose intolerance within the past 5 years. Apremilast pills contain lactose; however, the use of concurrent lactase enzyme in lactose intolerant participants will not be considered and lactose intolerant patients will still be excluded even if they take lactase enzyme supplementation. This is explained by the potential exacerbation of gastrointestinal symptoms with Apremilast as an Adverse Event (AE).
6. CYP3A4 inducers have been shown to diminish Apremilast levels (Lexi-Comp Online™ Interaction Monograph accessed August 1st, 2015); hence, patients will be excluded if they are on concomitant Carbamazepine, Enzalutamide, Fosphenytoin, Lumacaftor, Mitotane, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, and Rifapentine.
7. As per Celgene, the presence of any of the following will exclude a subject from enrollment:

   1. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
   2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
   3. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
   4. Pregnant or breast feeding.
   5. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
   6. Malignancy or history of malignancy, except for:

      * treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
      * treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
   7. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
   8. Prior treatment with apremilast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Assessing treatment success defined as Physician Global Assessment (PhGA) of 0 or 1 | Baseline to 16 weeks
  The primary outcome will be assessing treatment success with Apremilast as compared to placebo defined as Physician Global Assessment (PhGA) of 0 or 1.

SECONDARY OUTCOMES:
Achieving complete remission defined as achieving a score of 0 on PhGA scale | 12 weeks and 16 weeks
  Complete remission is defined as achieving a score of 0 on PhGA scale
Physician Global Assessment (PhGA) | Baseline to 16 weeks
  Physician Global Assessment (PhGA) grading score from 0 to 4. Score of 0 is clear, score of 1 is almost clear, score of 2 is mild disease, score of 3 is moderate disease, and a score of 4 is severe disease.
Patient Assessment (PtA) | Baseline to 16 weeks
  Patient Assessment (PtA) grading score from 0 to 4. Score of 0 is clear, score of 1 is almost clear, score of 2 is mild disease, score of 3 is moderate disease, and a score of 4 is severe disease.
Achieving partial response | Baseline to 12 weeks
  Percentage of patients who achieve partial response
Visual Analogue Scale (VAS) | Baseline to 16 weeks
  Patient assessment of pain score from 0 to 10. VAS is a scale demonstrated by a 10 cm horizontal line marked from 0-10 with the left end marked as no symptoms (0) and the right end marked as worst symptoms (10).
Oral Health Impact Profile (OHIP-14) Scale | Baseline to 16 weeks
  Patient assessment of overall disease impact on quality of life is a self-filled validated scale that focuses on seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Participants will be asked to respond according to frequency of impact on a 5-point scale coded: never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4).
Modified Oral Mucositis Index (MOMI) Scale | Baseline weeks to 16 weeks
  Physician assessment using a validated 20 item scale in OLP, is used to rate four types of mucosal changes (atrophy, edema, erythema, and ulceration) in nine anatomical areas of the oral cavity
Safety and tolerability of Apremilast | 6 weeks to 16 weeks
  Relationship of adverse events to study treatment. Difference in proportions between the two study arms for each AE at each time point will be assessed and changes in the incidence of treatment.
Standardized steroid and anti-fungal rinses used | 6 weeks to 16 weeks
  Differences in total dexamethasone and nystatin mouthwashes quantity used at each time point between the two study arms will be assessed
Body Mass Index (BMI) | Baseline to 16 weeks
  Differences in BMI scores at each time point between two study arms will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Klieb, HBSc, MSc, DMD, FRCD(C), Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No